CLINICAL TRIAL: NCT04192383
Title: Functional Magnetic Resonance Imaging Combined With Radiomics for Evaluation of Effectiveness of CyberKnife Stereotactic Radiosurgery for Spinal Tumors
Brief Title: Evaluation of Effectiveness of CyberKnife Stereotactic Radiosurgery for Spinal Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2018251
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-02

CONDITIONS: Spinal Neoplasms
Keywords: Spinal Neoplasms; Stereotactic Body Radiotherapy; CyberKnife Radiosurgery; Functional MRI; treatment outcome
MeSH Terms: conditions — Spinal Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cyberknife
  Interventions: Radiation: Cyberknife stereotactic radiosurgery

INTERVENTIONS:
Radiation: Cyberknife stereotactic radiosurgery — Hypofractionated stereotactic radiosurgery

SUMMARY:
This study aims to explore the reliability of the combination of functional magnetic resonance imaging and radiomics for evaluation of the therapeutic efficacy of CyberKnife stereotactic radiosurgery for spinal tumors. Accurate imaging assessment can help clinicians plan personalized therapeutic schedules for patients with spinal tumors .

DETAILED DESCRIPTION:
Spinal tumors may be metastases or primary tumors; the former are more common. About 40% of cancer patients will have spinal metastasis. Primary spinal tumor is relatively rare, accounting for only about 8% of spinal tumors. For both metastasis and primary tumor, the aim of treatment is to reduce pain, maintain or improve neurological function, and maintain or restore spinal stability.

In patients who cannot undergo surgery or need additional treatment after surgery, radiation therapy can relieve pain, prolong survival, improve the success rate of surgery, and reduce risk of metastasis and recurrence. However, the complex anatomy of the spine, and the numerous important organs around it, makes radiation treatment challenging. High-dose radiation therapy is necessary for long-term control of the tumor and for prevention of spinal column instability; however, this is impossible with traditional radiotherapy due to the presence of the radiosensitive spinal cord. Outcomes therefore tend to be poor for large and complex lesions. The CyberKnife-a stereotactic body radiation therapy (SBRT) platform that combines a lightweight linear accelerator, a robotic arm, an imaging system, and a respiratory tracking system-offers a feasible approach. It can achieve submillimeter level-precision treatment under imaging guidance.

Currently, the effectiveness of CyberKnife radiosurgery for spinal tumors is decided by assessing imaging changes, relief of clinical symptoms, and needle biopsy, but all of these methods have limitations. On imaging, for example, change in lesion volume is used to assess tumor regression, but the size of a spinal tumor is not easy to measure and, moreover, decrease in tumor volume after treatment may take time . Post-treatment signal intensity changes in conventional magnetic resonance imaging (MRI) T1-weighted and T2-weighted sequences are difficult to interpret, and their relationship with treatment efficacy is also not clear.

Generally speaking, alterations in microscopic structure and biological activity of the tumor occur much earlier than changes in gross morphology . Functional magnetic resonance imaging (fMRI) can therefore be more useful than conventional MRI for assessing treatment response. In fMRI, sequences such as diffusion-weighted imaging (DWI), dynamic contrast-enhanced MRI (DCE-MRI), and diffusion kurtosis imaging (DKI) reflect functional information of tissues from different perspectives.

Application of artificial intelligence technology for analysis of medical imaging data is now an area of intense research. This new method, which is called radiomics, can help in solving many difficult clinical problems. By extracting a large number of highly representative quantitative imaging features from high-throughput medical image data, radiomics can help in evaluating treatment efficacy and predicting prognosis of spinal tumors.

Investigators intend to explore the use of the combination of fMRI and radiomics for evaluating the effectiveness of CyberKnife radiosurgery for spinal tumors. The method will be able to evaluate both volume and functional changes in the tumor, and thus provide important information for planning of individualized therapeutic schedules for patients with spinal tumors.

ELIGIBILITY:
Inclusion criteria:

* Biopsy-proven spinal or paraspinal metastases;
* MRI and DCE-MRI examination performed before and at 3 months after CyberKnife treatment.

Exclusion criteria:

* Area of the lesion surgically removed before enrollment;
* Prior percutaneous vertebroplasty or kyphoplasty or radiation therapy of the target lesion;
* Chemotherapy within a month;
* Unable to cooperate with-or refusal of-CT, conventional MRI, or DCE-MRI examination;
* Lost to follow-up;
* Poor image quality that cannot be analyzed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohorts will be selected form Peking University Third Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | From the start of randomization to the date of death of the patient or the end of the study (at 60 months).
  The time from the start of treatment to the date of death or last follow-up

SECONDARY OUTCOMES:
Progression-free survival(PFS) | From the start of randomization to the first evidence of tumor progression or death of the patient or the end of the study (at 60 months), whichever occurs first.
  The time from the start of treatment to the date of diagnosis of tumor progression or death. Tumor progression is defined as increase in lesion volume on MRI compared to baseline, or identification of new metastasis on imaging or histological examination.
Numerical rating scales (NRS) | Measurements will be performed every 3 months, starting from randomization until the patient's death or till end of the study (at 60 months ).
  A 11 point scale where the end points are the extremes of no pain and pain as bad as it could be, or worst pain.
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Measurements will be performed every 3 months, starting from randomization until the patient's death or till end of the study (at 60 months ).
  The QLQ-C30 is a cancer-specific, self-administered, structured questionnaire designed for use in clinical trials, which contains 30 questions (items),

CONTACTS AND LOCATIONS:
Locations (1):
- Yongye Chen, Beijing, Beijing Municipality, China